CLINICAL TRIAL: NCT03671811
Title: Open-Label Randomized Phase II Trial of Megestrol Acetate With or Without Pterostilbene in Patients With Endometrial Cancer Scheduled for Hysterectomy
Brief Title: Megestrol Acetate With or Without Pterostilbene in Treating Patients With Endometrial Cancer Undergoing Hysterectomy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17327; NCI-2018-01555 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17327 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2018-07-27; First posted 2018-09-14 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Atypical Endometrial Hyperplasia; Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Megestrol Acetate; Pterocarpus marsupium; 3,5-dimethoxy-4'-hydroxystilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (pterostilbene, megestrol acetate) (Experimental): Patients receive 100mg pterostilbene BID and 80mg megestrol acetate PO BID for 3 weeks in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Megestrol Acetate; Biological: Pterostilbene
- Arm II (megestrol acetate) (Experimental): Patients receive megestrol acetate PO BID for 3 weeks in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Megestrol Acetate

INTERVENTIONS:
Drug: Megestrol Acetate — Given PO
  Other Names: 17-Hydroxy-6-methylpregna-4,6-diene-3,20-dione acetate; 17.alpha.-Acetoxy-6-methylpregna-4,6-diene-3,20-dione; 6-Dehydro-6-methyl-17.alpha.-acetoxyprogesterone; 6-Methyl-6-dehydro-17.alpha.-acetoxyprogesterone; BDH 1298; BDH-1298; Maygace; Megace; Megestat; Megestil; Niagestin; Ovaban; Pallace; SC-10363
Biological: Pterostilbene — Given PO
  Other Names: 3'',5''-Dimethoxy-4-stilbenol; 3,5-Dimethoxy-4''-hydroxystilbene; Trans-3,5-dimethoxy-4-hydroxystilbene
  Arms: Arm I (pterostilbene, megestrol acetate)

SUMMARY:
This phase II trial studies how well megestrol acetate with or without pterostilbene works in treating patients with endometrial cancer undergoing hysterectomy. Drugs used in chemotherapy, such as megestrol acetate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Pterostilbene is an antioxidant found in blueberries or grapes, and it has been shown to be effective in killing tumor cells and reducing cancer burden. It is not yet known whether giving megestrol acetate with or without pterostilbene may work better in treating patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of megestrol acetate (MA) plus pterostilbene (PTE) versus MA alone on tumor proliferation (Ki-67) during the preoperative window in patients with endometrial cancer (EC) who are scheduled for hysterectomy.

EXPLORATORY OBJECTIVES:

I. Determine the effect of MA plus PTE versus MA alone on histologic response during the preoperative window in patients with EC or endometrial complex atypical hyperplasia who are scheduled for hysterectomy.

II. Explore biological characteristics of tumors to determine potential biomarkers which could select for treatment eligibility in future studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pterostilbene orally (PO) twice daily (BID) and megestrol acetate PO BID for 3 weeks in the absence of disease progression or unaccepted toxicity.

ARM II: Patients receive megestrol acetate PO BID for 3 weeks in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Willing to undergo an intraoperative biopsy/or standard of care tissue collection during surgery, following completion of treatment with MA +/- PTE
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Histologically confirmed EC or complex atypical hyperplasia of the endometrium
* Candidate for a total hysterectomy with or without bilateral salpingo-oophorectomy
* About to initiate preoperative window period, with planned hysterectomy scheduled
* Platelets >= 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 1.5 x ULN
* Alanine aminotransferase (ALT) =< 1.5 x ULN
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Women of childbearing potential: negative urine or serum pregnancy test in premenopausal women. Postmenopausal women do not need to undergo a pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

Exclusion Criteria:

* Pterostilbene supplements within 30 days prior to day 1 of protocol therapy
* Any of the following phytochemical-based supplements within 30 days prior to day 1 of protocol therapy: resveratrol, genistein, and quercetin
* Chemotherapy for EC
* Allergic reaction/hypersensitivity to similar agents, excipients
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertensive emergency/urgency (defined as systolic blood pressure >= 180 mmHg and/or diastolic blood pressure >= 120 mmHg)
* Active or history of recent thromboembolism or stroke, within the past 6 months
* Cushing's syndrome
* Acute infection requiring systemic (intravenous) treatment
* Known history of human immunodeficiency virus (HIV) infection
* Known active hepatitis B or C infection
* Inability to swallow tablets/capsules
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2026-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh H Dellinger, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 patients were accrued. Seven patients were not evaluable for various reasons: received <10 days of study treatment (n = 5), disenrolled (n = 1), did not receive hysterectomy (n = 1). Consequently, 37 patients were randomized to treatment.
Period: Overall Study
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Started | 23 | 21
Completed | 19 | 18
Not Completed | 4 | 3
Not completed — Did not complete treatment (n=5), Disenrolled (n=1), Did not have hysterectomy (n=1) | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate) | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.3 [57.3 to 70.9] | 63.9 [56.7 to 71.5] | 61.9 [57.3 to 70.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 17 | 10 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Tumor Ki-67 Proliferation Index
Description: Ki-67 represents a specific nuclear marker for cell proliferation that is measured by staining with specific antibodies by immunohistochemical (IHC) staining. The Ki-67 proliferation index is defined as percent tumor cells staining positive, and measured on a continuous scale of 0-100%, with higher values indicating higher proliferation. Ki-67 hotspot values were assessed at two time-points during this study, prior to treatment with megace +/- pterostilbene (pre-treatment), and following completion of treatment (post-treatment). Descriptive statistics were used to compare treatment-associated percent change in Ki-67 proliferation index between the 2 study arms, using a 1-sided test with significance at p < 0.05.
Time Frame: Pre- and post-treatment up to 6 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 19 | 18
percent change | -26.7 (34.1) | -25.7 (36.3)
Statistical Analysis 1: Comparison: Arm I (Pterostilbene, Megestrol Acetate) vs Arm II (Megestrol Acetate); Test type: Superiority — The planned sample size was 36 evaluable participants, with 18 per treatment arm. Based on a one-sided t-test at α = 0.05, the study was designed to provide 90% power to detect a difference of at least 10 percentage points in the mean reduction of Ki-67 between arms, assuming a standard deviation of 10%. The difference was expected to favor the Pterostilbene + Megestrol Acetate arm; p = 0.9, t-test, 1 sided

2. Secondary Outcome: Histologic Response of Gland Cellularity
Description: These histologic changes represent measures of growth and apoptosis, and will be separately scored in the pretreatment endometrial sample and the section of tumor from the hysterectomy (post-treatment sample). Gland cellularity will be assessed by counting the number of cells in one quarter of a high-power field (HPF) (average of 3 fields). The number of patients with an improvement in gland cellularity were compared between study arms.
Time Frame: Up to 6 weeks
Population: Only 36 patients had data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 19 | 17
Participants | 13 | 14

3. Secondary Outcome: Histologic Response of Mitotic Index
Description: These histologic changes represent measures of growth and apoptosis, and will be separately scored in the pretreatment endometrial sample and the section of tumor from the hysterectomy (post-treatment sample). The mitotic index will be calculated as the number of mitoses per HPF (average of 3 fields). The number of patients with an improvement in mitotic index were compared between study arms.
Time Frame: Up to 6 weeks
Population: Only 36 patients had data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 19 | 17
Participants | 14 | 14

4. Secondary Outcome: Histologic Response of Metaplasia
Description: These histologic changes represent measures of growth and apoptosis, and will be separately scored in the pretreatment endometrial sample and the section of tumor from the hysterectomy (post-treatment sample). The percentages of tumor that display squamous or mucinous metaplasia will be estimated as percentages, with < 10% considered negative and >= 10% as positive. The number of patients with an improvement in metaplasia were compared between study arms.
Time Frame: Up to 6 weeks
Population: Only 36 patients had data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 19 | 17
Participants | 8 | 11

5. Secondary Outcome: Histologic Response of Eosinophilic Metaplasia
Description: These histologic changes represent measures of growth and apoptosis, and will be separately scored in the pretreatment endometrial sample and the section of tumor from the hysterectomy (post-treatment sample). The number of patients with an improvement in eosinophilic metaplasia were compared between study arms.
Time Frame: Up to 6 weeks
Population: Only 36 patients had data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 19 | 17
Participants | 9 | 5

6. Secondary Outcome: Immunohistochemical Expression of Bcl-2 to Assess Tumor Growth and Apoptosis
Description: Immunohistochemistry stains with antibodies directed against Bcl-2 will be performed on pre- and post-treatment endometrial samples. Samples will be scored on a continuous scale (0-100%) using the product of the intensity of cytoplasmic staining, and the proportion of cells staining based on the distribution of staining. Descriptive statistics were used to compare the percent change in scores from pre-treatment to post-treatment between the 2 study arms.
Time Frame: Pre- and post-treatment up to 6 weeks
Population: Only 33 patients had data for this endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 16 | 17
percent change | 2.1 (5.2) | 1.2 (4.4)
Statistical Analysis 1: Comparison: Arm I (Pterostilbene, Megestrol Acetate) vs Arm II (Megestrol Acetate); Test type: Superiority — This was a one-sided t-test at α = 0.05. The difference was expected to favor the Pterostilbene + Megestrol Acetate arm; p = 0.6, t-test, 1 sided

7. Secondary Outcome: Immunohistochemical Expression of Casp3 to Assess Tumor Growth and Apoptosis
Description: Immunohistochemistry stains with antibodies directed against Casp3 to assess apoptosis will be performed on pre- and post-treatment endometrial samples. Samples will be scored by counting the number of positive staining nuclei per HPF. Descriptive statistics were used to compare the percent change in scores from pre-treatment to post-treatment between the 2 study arms.
Time Frame: Pre- and post-treatment up to 6 weeks
Population: Only 25 patients had data for this endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
Number analyzed (Participants) | 13 | 12
percent change | -46.4 (48.7) | -8.8 (79.7)
Statistical Analysis 1: Comparison: Arm I (Pterostilbene, Megestrol Acetate) vs Arm II (Megestrol Acetate); Test type: Superiority — This was a one-sided t-test at α = 0.05. The difference was expected to favor the Pterostilbene + Megestrol Acetate arm; p = 0.2, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of surgery until the 6-week post-suregry visit.
Description: "Other Adverse Events" include all events that were not severe adverse events, regardless of grade or relation to treatment.
Arm/Group | Arm I (Pterostilbene, Megestrol Acetate) | Arm II (Megestrol Acetate)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 16/19 | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pterostilbene, Megestrol Acetate) (N=19) | Arm II (Megestrol Acetate) (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (6) | 4 (4)
Fever (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
cramping (General disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT03671811/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03671811/ICF_001.pdf